CLINICAL TRIAL: NCT06966089
Title: Evaluation of Urinary Exosomes as a Risk Stratification Tool Among Men With Elevated PSAs and Negative Prostate MRIs
Brief Title: ExosomeDx in MRI-negative Men With High PSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bio-Techne Corporation (Unknown)
Responsible Party: Principal Investigator, Nikhil Waingankar, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY-24-00010
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Urinary Exosome; ExoDx Prostate test; ExosomeDx; ERG; Erythroblast Transformation-Specific Related Gene; SPDEF; SAM Pointed Domain-containing ETS Transcription Factor; Exosome Diagnostic Intelligence; EPI; Prostate cancer; Prostate Biopsy; Exosome; Prostate MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective diagnostic test design will be used to compare the sensitivity of ExoDx with PSA density (H0: SensitivityPSA Density ≤ SensitivityExoDx versus H1: SensitivityPSA Density > SensitivityExoDx) and the specificity (H0: Specificity PSA Density ≤ Specificity ExoDxversus H1: Specificity PSA Density > Specificity ExoDx).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants with elevated or rising PSA (Experimental): Participants who have been diagnosed with an elevated or rising PSA as determined by their urologist, and who have a negative (PIRADS 1 or 2) prostate MRI will be offered enrollment in this trial. ExoDx Study Kit will be collected onsite. Participants will then be scheduled for transrectal ultrasound-guided or transperineal 12-core prostate biopsy as per the standard diagnostic practice.
  Interventions: Device: Urinary ExoDx test; Diagnostic Test: Transrectal ultrasound-guided prostate biopsy; Diagnostic Test: Transperineal 12-core prostate biopsy

INTERVENTIONS:
Device: Urinary ExoDx test — A urine sample for ExoDx Study Kit will be collected onsite and shipped to Exosome Diagnostic's laboratory.
Diagnostic Test: Transrectal ultrasound-guided prostate biopsy — Participants will be scheduled for transrectal ultrasound-guided prostate biopsy as per the standard diagnostic practice after urinary test.
Diagnostic Test: Transperineal 12-core prostate biopsy — Participants will be scheduled for transperineal 12-core prostate biopsy as per the standard diagnostic practice after urinary test.

SUMMARY:
Magnetic resonance imaging (MRI) has become the current standard of care in risk stratifying men with an elevated Prostate-specific antigen (PSA) to determine who needs to undergo prostate biopsy, which is invasive and carries a 3-5% risk of serious infection. Recent data shows the negative predictive value of MRI to be only 77%, indicating that some men may inappropriately forego biopsy based on a negative MRI. Urinary exosomes can be captured and analyzed by the ExosomeDx (ExoDx) Prostate test, a urine based, gene signature derived from PCA3 (prostate cancer antigen 3) and ERG (erythroblast transformation-specific related gene), and SPDEF (SAM pointed domain-containing ETS transcription factor); ExoDx carries a 90% negative predictive value.

The use of ExoDx test among patients with negative MRIs has the potential to improve the risk stratification of patients with an elevated PSA in a way that the Urologist can more accurately determine which patients need to undergo prostate biopsy. In doing so, the Urologist can better risk-stratify which patients should undergo prostate biopsy and be exposed to the associated potential risks, and also be more confident about the safety of foregoing biopsy in those patients with negative MRI and negative ExoDx test.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all the following criteria;

* Willingness to participate and provide signed and dated informed consent form
* Male (sex)
* Age ≥ 18 years
* PSA screen-eligible, per investigator discretion

  * 45-75 years of age for average risk
  * 40-75 years of age for high risk
* PSA ≥ 2.0 ng/mL and ≤ 10.0 ng/mL
* MRI PIRADS score of 1 or 2
* ECOG 0-1
* Must have a negative urine culture prior to biopsy
* No prior prostate biopsies within the last 5 years (biopsy-naïve)
* Willingness to undergo a prostate biopsy as part of the diagnostic work-up
* Digital rectal exam with no palpable nodules

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study;

* Prior or current histologic or pathologic confirmed diagnosis of prostate cancer
* Prior transrectal ultrasound within the last 5 years
* Any prior cancer diagnosis within the last 5 years
* On immunosuppression or predefined immunosuppressed state
* A known coagulopathy predisposition to bleeding
* Diagnoses of any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
* Cognitive inability or psychiatric conditions that preclude informed decision making or compliance with study requirements (per investigator discretion)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All men who present to Mount Sinai Health System urology clinic and, in the course of routine PSA screening, who are found to have an elevated PSA and a negative MRI (PIRADS 1 or 2) will be approached for consideration to participate in this study.
Enrollment: 425 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | duration of study, average 3 months
  Sensitivity is defined as the probability that clinically significant cancer is detected when it is cancer.
  Sensitivity = true positive cases / true positive cases + false negative cases
Specificity | duration of study, average 3 months
  Specificity is defined as the probability that clinically significant cancer is not detected when it is not cancer.
  Specificity = true negative cases / true negative cases + false positive cases

SECONDARY OUTCOMES:
Cancer Detection Rate | duration of study, average 3 months
  Cancer Detection Rate (CDR): Cancer detection rate is defined as the proportion of enrolled patients with histologically Gleason grade group 1+ cancers and as determined by the Investigator.
  Cancer detection rate = true positive (histologically Gleason grade 1+) / all tests performed
csPCa Detection Rate | duration of study, average 3 months
  csPCa Detection Rate (csCDR): clinically significant cancer detection rate is defined as the proportion of enrolled patients with histologically Gleason grade group 2+ cancers.
  csPCa detection rate = true positive (histologically Gleason grade 2+) / all tests performed
Biopsy aversion rate | duration of study, average 3 months
  Biopsy aversion rate is defined as the proportion of patients in whom the biopsy could have been potentially averted using ExosomeDx, as compared to decisions based on PSA density.
Net Benefit | duration of study, average 3 months
  Decision curve analysis will be used to calculate the net benefit of adding ExoDx to PSA density (including kinetics and density) and MRI in the diagnostic workflow following.
  Net benefit is calculated across a range of threshold probabilities, defined as the minimum probability of disease at which further intervention would be warranted, as net benefit = sensitivity × prevalence - (1 - specificity) × (1 - prevalence) × w where w is the odds at the threshold probability.
Diagnostic Accuracy | duration of study, average 3 months
  Accuracy is defined as the potential of ExoDx to correctly detect the presences or absence of disease.
  Diagnostic Accuracy = (True Positive) + True Negative / All) * 100
Positive Predictive Value (PPV) | duration of study, average 3 months
  Positive predictive value is defined as the probability that an elevated ExoDx actually has cancer.
  Positive Predictive Value = (True Positive)/(True Positive + False Positive)
Negative Predictive Value (NPV) | duration of study, average 3 months
  Negative predictive value is defined as the probability a negative ExoDx test does not cancer.
  Negative Predictive Value = (True Negative)/(True Negative + False Negative)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Waingankar, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (6):
- United States (6):
  - Mount Sinai Beth Israel / Union Square, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Morningside, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Mount Sinai Queens, New York, New York
  - Mount Sinai Brooklyn, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Specify Other Mechanism Email proposal to Principal Investigator.